CLINICAL TRIAL: NCT06257888
Title: The Journey of Women With Breast Cancer in Mozambique: What is the Best Path? A Prospective Cohort With Patient Navigation as an Intervention to Reduce Treatment Disparities
Brief Title: A Prospective Cohort With Patient Navigation as an Intervention for Breast Cancer Patients
Acronym: NAVIMOZ
Status: Completed | Type: Observational
Sponsor: Renato Cagnacci Neto (Other)
Collaborators: AMERICAN SOCIETY FOR CLINICAL PATHOLOGY (Unknown); Hospital Central de Maputo (Unknown); Eduardo Mondlane University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Renato Cagnacci Neto, Principal Investigator, AC Camargo Cancer Center
Organization: AC Camargo Cancer Center (Other)
Other Study IDs: CIBS FM&HCM/054/2023
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Malignant Primary
Keywords: breast cancer; malignant neoplasm of the breast; patient navigation; Carcinoma, Intraductal, Noninfiltrating
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Patient Navigation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- breast cancer patients under navigation: breast cancer patients, intervention = patient navigation
  Interventions: Other: patient navigation

INTERVENTIONS:
Other: patient navigation — two trained patient navigators will admit breast cancer patients to HCM, navigate them from admission to commencement of first treatment and will collect all pertinent epidemiological data and variables

SUMMARY:
The objective of this observational study is to introduce a patient navigation system within the breast cancer unit at Hospital Central de Maputo (MOZ) and gather data to assess the efficacy of patient navigation in enhancing oncological outcomes among this patient cohort. The primary inquiries it seeks to address are as follows:

* Can patient navigation reduce the duration (in days) between patient admission and the commencement of treatment?
* Does patient navigation influence overall survival rates when juxtaposed with historical cohorts from the local setting? Participants will receive continuous support from a patient navigator starting from admission until the initiation of any oncological treatment.

DETAILED DESCRIPTION:
-General Objective: To implement an oncological navigation platform for breast cancer patients receiving treatment at Maputo Central Hospital (HCM) over a proposed period of 12 months after project approval by the local IRB.

-Specific Objectives:

* Develop an oncological patient navigation system for breast cancer patients treated at HCM.
* Establish a prospective cohort of navigated breast cancer patients (with invasive or ductal carcinoma in situ) treated at HCM in 2024-25 (recruitment period of twelve months).
* Collect diverse epidemiological data from navigated patients during the proposed study period.
* Describe the following variables: time from first symptom until first medical consultation (in days), time from first medical consultation to cancer diagnosis (in days) and time from diagnosis to first treatment (either surgery or neoadjuvant treatment) in days.
* Compare time from first symptom to diagnosis (in days) and time from diagnosis to first treatment (in days) to a historical cohort published by Brandão M. et al (The Oncologist, 2021).
* Collect overall survival data in this cohort for thirty six months after last patient recruited for future publication.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 years and older
* will undergo breast cancer treatment at HCM
* consent to participate

Exclusion Criteria:

* male
* less than18 years of age
* history of other previous malignancies (including breast cancer)
* history of breast cancer treatment initiated elsewhere
* lack of consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: we will recruit all female primary breast cancer patients (invasive or in situ) admitted for treatment at HCM during a 12 month period
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
time interval between first symptom and first medical consultation | 12 months
  time interval (in days) between first symptom and first medical consultation (either at Maputo Central Hospital or any other medical service)
time interval between first medical consultation and cancer diagnosis | 12 months
  time interval (in days) between first medical consultation (at Maputo Central Hospital) and cancer diagnosis (by any type of biopsy performed at Maputo Central Hospital)
time interval between cancer diagnosis and first treatment | 12 months
  time interval (in days) between cancer diagnosis (by any type of biopsy performed at Maputo Central Hospital) and first treatment (surgery or neoadjuvant chemotherapy at Maputo Central Hospital)
overall survival | 36 months after last patient recruited
  overall survival (in months) of navigated breast cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: renato cagnacci neto, MD, MSc, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- Hospital Central de Maputo, Maputo, Cidade de Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
we will share all collected IPD with any researchers that contact the PI
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: available after publication for one year

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Lorenzoni CF, Ferro J, Carrilho C, Colombet M, Parkin DM. Cancer in Mozambique: Results from two population-based cancer registries. Int J Cancer. 2020 Sep 15;147(6):1629-1637. doi: 10.1002/ijc.32953. Epub 2020 Mar 18. PMID 32142162
- [Background] Brandao M, Guisseve A, Bata G, Firmino-Machado J, Alberto M, Ferro J, Garcia C, Zaqueu C, Jamisse A, Lorenzoni C, Piccart-Gebhart M, Leitao D, Come J, Soares O, Gudo-Morais A, Schmitt F, Tulsidas S, Carrilho C, Lunet N. Survival Impact and Cost-Effectiveness of a Multidisciplinary Tumor Board for Breast Cancer in Mozambique, Sub-Saharan Africa. Oncologist. 2021 Jun;26(6):e996-e1008. doi: 10.1002/onco.13643. Epub 2021 Jan 6. PMID 33325595
- [Background] Rosa DD, Bines J, Werutsky G, Barrios CH, Cronemberger E, Queiroz GS, de Lima VCC, Freitas-Junior R, Couto JD, Emerenciano K, Resende H, Crocamo S, Reinert T, Van Eyil B, Neron Y, Dybal V, Lazaretti N, de Cassia Costamilan R, de Andrade DAP, Mathias C, Vacaro GZ, Borges G, Morelle A, Caleffi M, Filho CS, Mano MS, Zaffaroni F, de Jesus RG, Simon SD. The impact of sociodemographic factors and health insurance coverage in the diagnosis and clinicopathological characteristics of breast cancer in Brazil: AMAZONA III study (GBECAM 0115). Breast Cancer Res Treat. 2020 Oct;183(3):749-757. doi: 10.1007/s10549-020-05831-y. Epub 2020 Jul 29. PMID 32728860
- [Background] Simon SD, Bines J, Werutsky G, Nunes JS, Pacheco FC, Segalla JG, Gomes AJS, Adam Van Eyll BMHR, Gimenes DL, Crocamo S, Freitas-Junior R, Lago LD, Queiroz GS, Jobim de Azevedo S, Rosa DD, Delgado G, Borges GS, Veronica do Nascimento Y, Zaffaroni F, Martinez-Mesa J, Barrios CHE. Characteristics and prognosis of stage I-III breast cancer subtypes in Brazil: The AMAZONA retrospective cohort study. Breast. 2019 Apr;44:113-119. doi: 10.1016/j.breast.2019.01.008. Epub 2019 Feb 2. PMID 30738289
- [Background] Tulsidas S, Fontes F, Brandao M, Lunet N, Carrilho C. Oncology in Mozambique: Overview of the Diagnostic, Treatment, and Research Capacity. Cancers (Basel). 2023 Feb 11;15(4):1163. doi: 10.3390/cancers15041163. PMID 36831505
- [Background] Budde H, Williams GA, Scarpetti G, Kroezen M, Maier CB. What are patient navigators and how can they improve integration of care? [Internet]. Copenhagen (Denmark): European Observatory on Health Systems and Policies; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK577640/ PMID 35129934
- [Background] Ramirez A, Perez-Stable E, Penedo F, Talavera G, Carrillo JE, Fernandez M, Holden A, Munoz E, San Miguel S, Gallion K. Reducing time-to-treatment in underserved Latinas with breast cancer: the Six Cities Study. Cancer. 2014 Mar 1;120(5):752-60. doi: 10.1002/cncr.28450. Epub 2013 Nov 12. PMID 24222098
- [Background] Raj A, Ko N, Battaglia TA, Chabner BA, Moy B. Patient navigation for underserved patients diagnosed with breast cancer. Oncologist. 2012;17(8):1027-31. doi: 10.1634/theoncologist.2012-0191. Epub 2012 Jul 2. PMID 22752069
- [Background] Cacala SR, Farrow H, Makhanya S, Couch DG, Joffe M, Stopforth L. The Value of Navigators in Breast Cancer Management in a South African Hospital. World J Surg. 2021 May;45(5):1316-1322. doi: 10.1007/s00268-020-05931-2. Epub 2021 Jan 18. PMID 33462702
- [Background] Rodrigues RL, Schneider F, Kalinke LP, Kempfer SS, Backes VMS. Clinical outcomes of patient navigation performed by nurses in the oncology setting: an integrative review. Rev Bras Enferm. 2021 Apr 16;74(2):e20190804. doi: 10.1590/0034-7167-2019-0804. eCollection 2021. English, Portuguese. PMID 33886831
- [Background] Koffi KG, Silue DA, Laurent C, Boidy K, Koui S, Compaci G, Adeba ZH, Kamara I, Botty RP, Bognini AS, Sanogo I, Despas F, Laurent G. AMAFRICA, a patient-navigator program for accompanying lymphoma patients during chemotherapy in Ivory Coast: a prospective randomized study. BMC Cancer. 2019 Dec 23;19(1):1247. doi: 10.1186/s12885-019-6478-3. PMID 31870438
- [Background] Chidebe RCW, Pratt-Chapman ML. Oncology Patient Navigation Training: Results of a Pilot Study in Nigeria. J Cancer Educ. 2022 Aug;37(4):1172-1178. doi: 10.1007/s13187-020-01935-7. Epub 2021 Jan 7. PMID 33411251
- [Background] Henderson V, Tossas-Milligan K, Martinez E, Williams B, Torres P, Mannan N, Green L, Thompson B, Winn R, Watson KS. Implementation of an integrated framework for a breast cancer screening and navigation program for women from underresourced communities. Cancer. 2020 May 15;126 Suppl 10:2481-2493. doi: 10.1002/cncr.32843. PMID 32348565